CLINICAL TRIAL: NCT02659540
Title: A Pilot (Phase 1) Study to Evaluate the Safety and Efficacy of Combination Checkpoint Blockade (Ipilimumab and Nivolumab) Plus External Beam Radiotherapy in Subjects With Stage IV Melanoma
Brief Title: Pilot Study of the Safety/Efficacy of Combination Checkpoint Blockade + External Beam Radiotherapy in Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Bristol-Myers Squibb (Industry); Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2015-006
Record Dates: First submitted 2016-01-06; First posted 2016-01-20 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Ipilimumab; Nivolumab; Radiotherapy
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Conventional RT) (Experimental): Subjects received concurrent ipilimumab (3 mg/kg) and nivolumab (1 mg/kg) every 3 weeks for 4 doses (i.e., Weeks 1, 4, 7 and 10), followed by nivolumab monotherapy administered at a dose of 240 mg every 2 weeks through Week 18. Continued nivolumab monotherapy was permitted beyond Week 18 at the Investigator's discretion as either 240 mg every 2 weeks or 480 mg every 4 weeks starting at Week 20. Extracranial RT was initiated after the first dose and before the second dose of immunotherapy and was administered to a target lesion at a conventional total palliative dose of 30 Gy delivered over 2 weeks in 10 fractions of 3 Gy each.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiotherapy
- Cohort B (Hypofractionated RT) (Experimental): Subjects received concurrent ipilimumab (3 mg/kg) and nivolumab (1 mg/kg) every 3 weeks for 4 doses (i.e., Weeks 1, 4, 7 and 10), followed by nivolumab monotherapy administered at a dose of 240 mg every 2 weeks through Week 18. Continued nivolumab monotherapy was permitted beyond Week 18 at the Investigator's discretion as either 240 mg every 2 weeks or 480 mg every 4 weeks starting at Week 20. Extracranial RT was initiated after the first dose and before the second dose of immunotherapy and was administered to a target lesion at a hypofractionated high-dose of 27 Gy delivered over 2 weeks in 3 fractions of 9 Gy each.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab was administered as an intravenous (IV) infusion over approximately 30 or 90 minutes, with dosing calculated using body weight.
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab was administered as an IV infusion over approximately 30 or 90 minutes, with dosing calculated using body weight. The ipilimumab infusion was initiated approximately 30 minutes after the end of the nivolumab infusion on applicable dosing days.
  Other Names: Yervoy
Radiation: Radiotherapy — RT was delivered in accordance with cohort assignment and institutional practices.

SUMMARY:
This is an ongoing, Phase 1, open-label, multicenter, pilot study of the checkpoint antibodies ipilimumab and nivolumab in combination with radiotherapy (RT) in 18 subjects with unresectable Stage IV melanoma. The primary study objective is to evaluate the safety of study treatment. Secondary objectives are to evaluate objective response rate (ORR) and disease control rate (DCR) at Weeks 12 and 18, duration of response, progression-free survival (PFS), and overall survival (OS).

DETAILED DESCRIPTION:
All subjects received concurrent ipilimumab (3 mg/kg) and nivolumab (1 mg/kg) every 3 weeks for 4 doses (i.e., Weeks 1, 4, 7 and 10), followed by nivolumab monotherapy administered at a dose of 240 mg every 2 weeks through Week 18. Continued nivolumab monotherapy was permitted beyond Week 18 at the Investigator's discretion as either 240 mg every 2 weeks or 480 mg every 4 weeks starting at Week 20. Extracranial RT was initiated after the first dose and before the second dose of immunotherapy, with RT dosing administered to a target lesion as follows:

* Cohort A: conventional total palliative dose of 30 Gy delivered over 2 weeks in 10 fractions of 3 Gy each;
* Cohort B: hypofractionated high-dose of 27 Gy delivered over 2 weeks in 3 fractions of 9 Gy each.

Eligible subjects were initially enrolled into Cohort A. After 9 evaluable subjects completed at least the first 2 cycles of concurrent ipilimumab and nivolumab treatment, a safety review was performed and determined that the safety of Cohort A was acceptable based on a protocol-specified tolerability threshold of ≤ 7 of 9 subjects experiencing Grade 3 or 4 drug- or radiation-related adverse events (AEs), where Grade 3 or 4 amylase or lipase abnormalities that were not associated with clinical symptoms were not included in the safety assessment. Additional subjects were then accrued to Cohort B.

Subjects were followed on study for 100 days after the last study drug administration. Post-study follow-up, which occurs at least every 12 (± 1) weeks for 3 years after completion of the 100-day on-study follow-up, is still being performed for some patients .

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of Stage IV metastatic melanoma, with 1 melanoma lesion that could be safely irradiated and, in the opinion of the radiation oncologist, was of benefit to the subject to irradiate (note: subjects with primary ocular and mucosal melanoma were permitted). Lesions may have included, but were not limited to:

   1. Symptomatic lymphadenopathy;
   2. Bothersome cutaneous disease;
   3. Hepatic metastases;
   4. Pulmonary metastases.
2. Excluding the lesion intended to undergo radiation, subjects must have had at least 1 unresectable, non-bony lesion that was measurable radiographically (based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
3. Any number of prior therapies (including none). For subjects who had received prior systemic treatment with cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4), programmed cell death-1 (PD-1), and/or programmed cell death ligand-1 (PD-L1) therapy, the last monoclonal antibody administration should have been no less than 4 weeks prior to start of this protocol therapy and all prior side effects must have resolved to grade 1 or less by the time of the start of this protocol therapy.
4. Subjects must have:

   * Completed investigational therapy, other immunotherapy, or prior RT at least 28 days before administration of the first dose of study drug(s)
   * Completed chemotherapy or targeted therapy at least 14 days before administration of the first dose of study drug(s)
   * Sufficiently recovered from prior surgery as determined by the treating Investigator.

   Clinically significant toxicity or pharmacodynamic effects experienced during any prior therapy must have been resolved or stabilized before the first dose of study drug(s).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Life expectancy ≥ 4 months.
7. Screening laboratory parameters:

   1. White blood cell count ≥ 2000/μL;
   2. Absolute neutrophil count ≥ 1500/μL;
   3. Platelets ≥ 100,000/μL;
   4. Hemoglobin ≥ 9 g/dL;
   5. Aspartate aminotransferase and alanine aminotransferase ≤ 3 × upper limit of normal (ULN);
   6. Total bilirubin ≤ 1.5 × ULN (< 3 mg/dL for subjects with Gilbert's disease);
   7. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

      * Female CrCl = [(140 - age in years) x weight in kg x 0.85] / [72 x serum creatinine in mg/dL];
      * Male CrCl = [(140 - age in years) x weight in kg x 1.00] / [72 x serum creatinine in mg/dL].
8. Age ≥ 18 years.
9. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Unresolved immune-related AEs following prior biological therapy. Subjects with asymptomatic endocrinopathy may have enrolled.
2. Active autoimmune disease or any condition requiring systemic treatment with either corticosteroids (>10 mg daily of prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents were permitted in the absence of active autoimmune disease.
3. History of motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre Syndrome, Myasthenia Gravis).
4. Other active, concurrent malignancy that required ongoing systemic treatment or interfered with radiographic assessment of melanoma response as determined by the Investigator.
5. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases were eligible if metastases had been treated and there was no magnetic resonance imaging (MRI) evidence of progression for 4 weeks or more after treatment was completed and within 28 days prior to the first dose of nivolumab administration. There must also have been no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
6. Known immunodeficiency or human immunodeficiency virus, Hepatitis B, or Hepatitis C positivity. Antibody to Hepatitis B or C without evidence of active infection may have been allowed.
7. History of severe allergic reactions to any unknown allergens or any components of the study drugs.
8. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
9. Requirement of RT to treat brain metastases or receipt of any non-study systemic therapy for cancer or any other experimental/investigational treatment.
10. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
11. Lack of availability for immunological and clinical assessments or post-study follow-up contact to determine relapse and survival.
12. Women who were breastfeeding or who were pregnant as evidenced by a positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) performed within 14 days of the first dose of study drug and by a urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours of the first dose of study drug(s).
13. Females of childbearing potential who were sexually active with a nonsterilized male partner must have used 2 methods of effective contraception from screening, and must have agreed to continue using such precautions for 23 weeks after the final dose of investigational product; cessation of birth control after this point should have been discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

    [Females of childbearing potential were defined as those who were not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).] Nonsterilized males who were sexually active with a female partner of childbearing potential must have used 2 acceptable methods of effective contraception from Day 1 and for 31 weeks after receipt of the final dose of investigational product.
14. Any condition that, in the clinical judgment of the treating physician, was likely to interfere with the interpretability of the data or prevent the subject from complying with any aspect of the protocol or that may have put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Postow, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Stanford Cancer Institute, Stanford, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST. Ann Oncol. 2014;25(Supplement 4):iv361-iv72.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Conventional RT): Subjects received concurrent ipilimumab (3 mg/kg IV) and nivolumab (1 mg/kg IV) every 3 weeks for 4 doses (i.e., Weeks 1, 4, 7 and 10), followed by nivolumab monotherapy administered at a dose of 240 mg IV every 2 weeks through Week 18. Continued nivolumab monotherapy was permitted beyond Week 18 at the Investigator's discretion as either 240 mg IV every 2 weeks or 480 mg IV every 4 weeks starting at Week 20. Extracranial RT was initiated after the first dose and before the second dose of immunotherapy and was administered to a target lesion at a conventional total palliative dose of 30 Gy delivered over 2 weeks in 10 fractions of 3 Gy each.
- Cohort B (Hypofractionated RT): Subjects received concurrent ipilimumab (3 mg/kg IV) and nivolumab (1 mg/kg IV) every 3 weeks for 4 doses (i.e., Weeks 1, 4, 7 and 10), followed by nivolumab monotherapy administered at a dose of 240 mg IV every 2 weeks through Week 18. Continued nivolumab monotherapy was permitted beyond Week 18 at the Investigator's discretion as either 240 mg IV every 2 weeks or 480 mg IV every 4 weeks starting at Week 20. Extracranial RT was initiated after the first dose and before the second dose of immunotherapy and was administered to a target lesion at a hypofractionated high-dose of 27 Gy delivered over 2 weeks in 3 fractions of 9 Gy each.
Period: Overall Study
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Started | 10 | 10
Completed (Completed treatment through Week 18) | 4 | 2
Not Completed | 6 | 8
Not completed — Adverse Event | 3 | 2
Not completed — Death | 1 | 0
Not completed — Progressive disease | 2 | 6

BASELINE CHARACTERISTICS:
Population: The population comprises all subjects who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [28 to 86] | 51 [37 to 76] | 60 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    0 | 4 | 5 | 9
    1 | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) were reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent was signed through 100 days after the last dose of study treatment. Treatment-emergent AEs were those that occurred or worsened after administration of the first dose of study treatment.
Time Frame: Up to 25 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
Participants
  Any TEAE | 10 | 10
  Treatment-related TEAE | 10 | 10
  Serious TEAE | 6 | 5

2. Secondary Outcome: Number of Subjects With Tumor Response at Week 12 by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at Weeks 12, 18, and 24, and every 12 weeks (± 7 days) thereafter until progression or start of alternate anticancer therapy. Per RECIST 1.1, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria (Eisenhauer et al. Eur J Cancer 2009;45:228-47).
Time Frame: 12 weeks
Population: The population comprises all subjects who received at least one dose of study treatment and had a Week 12 imaging assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
Participants
  PR | 4 | 0
  SD | 1 | 3
  PD | 5 | 6
  Not evaluated | 0 | 1

3. Secondary Outcome: Number of Subjects With Tumor Response at Week 18 by RECIST 1.1
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at Weeks 12, 18, and 24, and every 12 weeks (± 7 days) thereafter until progression or start of alternate anticancer therapy. Per RECIST 1.1, target lesions are categorized as follows: CR: Disappearance of all target lesions; PR: ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions; SD: small changes that do not meet above criteria (Eisenhauer et al. Eur J Cancer 2009;45:228-47).
Time Frame: 18 weeks
Population: The population comprises all subjects who received at least one dose of study treatment and had a Week 18 imaging assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
Participants
  PR | 4 | 0
  SD | 1 | 2
  PD | 5 | 7
  Not evaluated | 0 | 1

4. Secondary Outcome: Number of Subjects With Tumor Response at Week 12 by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at Weeks 12, 18, and 24, and every 12 weeks (± 7 days) thereafter until progression or start of alternate anticancer therapy. Per irRECIST, measurable lesions are categorized as follows: irCR: Complete disappearance of all target lesions; irPR: ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); irPD: ≥ 20% increase from nadir in TMTB; irSD: not meeting above criteria (Bohnsack et al. Ann Oncol 2014;25: iv361-iv72).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
Participants
  irPR | 4 | 0
  irSD | 1 | 3
  irPD | 5 | 6
  Not evaluated | 0 | 1

5. Secondary Outcome: Number of Subjects With Tumor Response at Week 18 by irRECIST
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at Weeks 12, 18, and 24, and every 12 weeks (± 7 days) thereafter until progression or start of alternate anticancer therapy. Per irRECIST, measurable lesions are categorized as follows: irCR: Complete disappearance of all target lesions; irPR: ≥ 30% decrease from baseline in the TMTB; irPD: ≥ 20% increase from nadir in TMTB; irSD: not meeting above criteria (Bohnsack et al. Ann Oncol 2014;25: iv361-iv72).
Time Frame: 18 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
Participants
  irPR | 4 | 0
  irSD | 1 | 2
  irPD | 5 | 7
  Not evaluated | 0 | 1

6. Secondary Outcome: Duration of Response
Description: Duration of response will be determined for each subject with time origin at the first occurrence of response until the first occurrence of progression or date of death if the subject dies due to any causes before progression. Every effort will be made to follow subjects for progression after they discontinue the study.
Time Frame: Up to 3 years post-study
Population: Duration of response was not measured in this study
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent of Patients With Progression-free Survival at 3 and 6 Months Post Start of Treatment
Description: Progression-free survival will be defined as the number of days from the date of first dose of study drug to the date of earliest disease progression or to the date of death, if disease progression does not occur. Subjects who do not progress and are still alive will be censored on the date of last follow-up or start of new treatment, whichever comes first. Living patients were censored at last off-study follow-up visit, last scan date, or at the end of study if no follow-up was available. PFS was estimated by Kaplan-Meier methodology.
Time Frame: At 3 and 6 months after the start of treatment
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
percent of participants
  Progression-free Survival at 3 months | 50 [18.4 to 75.3] | 50 [18.4 to 75.3]
  Progression-free Survival at 6 months | 50 [18.4 to 75.3] | 20 [3.1 to 47.5]

8. Secondary Outcome: Percent of Patients With Overall Survival at 12 Months Post Start of Treatment
Description: Overall survival (OS) will be measured for each subject from the date of the first dose of study drug until the recorded date of death or last follow-up. Subjects who are still alive will be censored on the date of last follow-up. Living patients were censored at last off-study follow-up visit, last scan date, or at the end of study if no follow-up was available. OS were estimated by Kaplan-Meier methodology.
Time Frame: Up to 12 months
Population: The population comprises all subjects who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
Number analyzed (Participants) | 10 | 10
percent of participants | 56.3 [20.9 to 80.9] | 56.3 [20.9 to 80.9]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date (i.e., through 100 days after the last dose of study treatment) were documented, regardless of the causal relationship to study drug. AEs that occurred or worsened in severity after the first dose of study treatment were considered treatment emergent (i.e., TEAEs).
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Cohort A (Conventional RT) | Cohort B (Hypofractionated RT)
All-Cause Mortality (participants affected / at risk) | 4/10 | 5/10
Serious Adverse Events (participants affected / at risk) | 6/10 | 5/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Conventional RT) (N=10) | Cohort B (Hypofractionated RT) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Suprapubic pain (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Anorectal infection (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Conventional RT) (N=10) | Cohort B (Hypofractionated RT) (N=10)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 2 | 1
Face oedema (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 7 | 6
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Mass (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 4 | 2
Pyrexia (General disorders) | 3 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Lipase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 3
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperactive pharyngeal reflex (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 2
Mucosal infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Palpitations (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 3 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Hypophysitis (Endocrine disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Wound drainage (Surgical and medical procedures) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Weight increased (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT02659540/Prot_SAP_000.pdf